CLINICAL TRIAL: NCT04896385
Title: A Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Mechanism of Action of Ruxolitinib Cream for Vitiligo
Brief Title: A Study to Evaluate the Mechanism of Action of Ruxolitinib Cream in Subjects With Vitiligo (TRuE-V MOA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-214; 2021-000361-32 (EudraCT Number)
Record Dates: First submitted 2021-04-30; First posted 2021-05-21 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
Keywords: Vitiligo; depigmenting disorder; topical JAK inhibitor
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, vehicle-controlled, with an open-label treatment extension.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib cream (Experimental): Ruxolitinib cream will be administered twice a day (BID) for 24 weeks
  Interventions: Drug: Ruxolitinib cream
- Vehicle Cream (Placebo Comparator): Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
  Arms: Ruxolitinib cream
Drug: Vehicle Cream — Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.
  Other Names: Placebo
  Arms: Vehicle Cream

SUMMARY:
The purpose of the study is to evaluate the Mechanism Of Action (MOA) of ruxolitinib cream in vitiligo by assessing the change in biomarkers.

ELIGIBILITY:
Inclusion Criteria

* A clinical diagnosis of nonsegmental vitiligo with depigmented areas including ≥ 0.5% BSA on the face, ≥ 0.5 F-VASI, ≥ 3% BSA on nonfacial areas, and ≥ 3 T-VASI; total body vitiligo area (facial and nonfacial) should not exceed 50% BSA.
* At least 1 active vitiligo lesion (eg, such as confetti lesion, trichrome appearance, pinkish rim, or other evidence of inflammatory activity) at the site for skin biopsy.
* Agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit. Over-the-counter preparations deemed acceptable by the investigator and camouflage makeups are permitted.

Exclusion Criteria

* No pigmented hair within any of the vitiligo areas on the face.
* Other forms of vitiligo (eg, segmental) or other differential diagnosis of vitiligo or other skin depigmentation disorders (eg, piebaldism, pityriasis alba, leprosy, postinflammatory hypopigmentation, progressive macule hypomelanosis, nevus anemicus, chemical leukoderma, and tinea versicolor).
* Used depigmentation treatments (eg, monobenzone) for past treatment of vitiligo or other pigmented areas except hydroquinone.
* Any other skin disease that, in the opinion of the investigator, would interfere with the study medication application or study assessments.
* Conditions at baseline that would interfere with evaluation of vitiligo.
* Use of any protocol-defined treatments within the indicated washout period before baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - First Oc Dermatology, Fountain Valley, California
  - UC Irvine, Irvine, California
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Suny Downstate Medical Center, Brooklyn, New York
  - Mount Sinai Hospital, New York, New York
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (4):
  - Dermatology Research Institute, Calgary, Alberta
  - Simcoderm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - JRB Research Inc, Ottawa, Ontario
- France (3):
  - Hopital Saint Andre, Bordeaux
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Archet 2 Derm Dept, Nice

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at a total of 11 sites in Canada, France, and the United States.
Groups:
- Double-Blind Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 24 weeks.
- Double-Blind Period: Vehicle Cream BID: Participants applied matching vehicle cream BID for 24 weeks.
- Treatment-Extension Period: Ruxolitinib Cream 1.5% BID: Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 28 weeks in the Treatment-Extension Period.
- Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID: Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5% BID for 28 weeks in the Treatment-Extension Period.
Period: 24-Week Double-Blind Period
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 41 | 19 | 0 | 0
Completed | 37 | 14 | 0 | 0
Not Completed | 4 | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Period: 28-Week Treatment-Extension Period
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 0 | 0 | 37 | 14
Completed | 0 | 0 | 27 | 9
Not Completed | 0 | 0 | 10 | 5
Not completed — Lost to Follow-up | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Participant Refused Safety Follow-up | 0 | 0 | 3 | 2
Not completed — Pregnancy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Total
Number analyzed (Participants) | 41 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.73) | 43.7 (13.16) | 44.7 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 26
  Male | 23 | 11 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 30 | 14 | 44
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 25 | 13 | 38
  Black/African-American | 4 | 2 | 6
  Asian | 5 | 3 | 8
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  Not Reported | 5 | 0 | 5
  South Asian | 1 | 0 | 1
  Middle Eastern | 0 | 1 | 1
Chemokine (C-X-C Motif) Ligand 10 (CXCL10), an immune biomarker [Mean (Standard Deviation); unit: nanograms per Liter (ng/L)] — Baseline was defined as the last non-missing measurement obtained on or before the first application of study drug. Population: Only participants with available data were analyzed.
  nanograms per Liter (ng/L)
    number analyzed (Participants) | 40 | 18 | 58
    (all) | 600.066 (959.3097) | 415.471 (177.4902) | 542.778 (804.0389)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Chemokine (C-X-C Motif) Ligand 10 (CXCL10), an Immune Biomarker, at Week 4, Week 12, and Week 24
Description: Baseline was defined as the last non-missing measurement obtained on or before the first application of study drug. Percentage change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value)*100.
Time Frame: Baseline; Week 4, Week 12, and Week 24
Population: Safety Population: all participants who applied at least 1 dose of study drug. Treatment groups for this population were to be determined according to the actual treatment the participant received on Day 1. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 39 | 16 | 0 | 0
percent change
  Week 4 | -20.93 (36.216) | 8.13 (52.491) |  |
  Week 12: number analyzed (Participants) | 37 | 14 | 0 | 0
  Week 12 | -18.33 (40.035) | 21.13 (70.690) |  |
  Week 24: number analyzed (Participants) | 35 | 14 | 0 | 0
  Week 24 | -12.92 (46.146) | 22.17 (68.893) |  |

2. Secondary Outcome: Correlation of Key Skin Inflammatory Biomarkers of Vitiligo in Target Lesions to Efficacy Readouts
Description: Clinical scores (facial Vitiligo Area Scoring Index [F-VASI] and total body Vitiligo Area Scoring Index [T-VASI]) were evaluated for correlation with skin CXCL10 levels.
Time Frame: Baseline, Week 12, and Week 24
Population: Safety Population. Repeated measures correlation (Crm) takes into account that measures were taken from the same individual across multiple timepoints. Included in the analysis were only those participants with values at each of 3 timepoints: Baseline, Week 12, and Week 24.
Measure: Number; unit: correlation coefficient
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 38 | 17
correlation coefficient
  F-VASI | -0.34 | 0.15
  T-VASI | -0.43 | 0.02
Statistical Analysis 1: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID; F-VASI; Test type: Other; p = 0.004, repeated measures correlation
Statistical Analysis 2: Comparison: Double-Blind Period: Vehicle Cream BID; F-VASI; Test type: Other; p = 0.41, repeated measures correlation
Statistical Analysis 3: Comparison: Double-Blind Period: Ruxolitinib Cream 1.5% BID; T-VASI; Test type: Other; p = 0.0002, repeated measures correlation
Statistical Analysis 4: Comparison: Double-Blind Period: Vehicle Cream BID; T-VASI; Test type: Other; p = 0.91, repeated measures correlation

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Double-Blind Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from the time of Informed Consent Form signing until the start of the Treatment-Extension Period or 30 days after the last application of study drug during the Double-Blind Period (up to Week 24 + 30 days)
Population: Double-Blind Safety Population: all participants who applied ruxolitinib cream or vehicle cream at least once during the Double-Blind Period. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 41 | 19
Participants | 19 | 7

4. Secondary Outcome: Number of Participants With TEAEs During the Treatment-Extension Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from the completion of the Week 24 assessments until at least 30 days after the last application of study drug at Week 52 + 30 days
Population: Treatment-Extension Evaluable Population: all participants who applied ruxolitinib cream at least once during the Treatment-Extension Period
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 37 | 14
Participants | 12 | 3

5. Secondary Outcome: Number of Participants With a Grade 3 or Higher TEAE During the Double-Blind Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. AE severity was assessed per the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated; Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living; Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: life-threatening consequences; urgent treatment indicated; Grade 5: fatal.
Time Frame: as for outcome 3
Population: Double-Blind Safety Population. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period: Ruxolitinib Cream 1.5% BID | Double-Blind Period: Vehicle Cream BID
Number analyzed (Participants) | 41 | 19
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With a Grade 3 or Higher TEAE During the Treatment-Extension Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. AE severity was assessed per the CTCAE, version 5.0: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated; Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living; Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: life-threatening consequences; urgent treatment indicated; Grade 5: fatal.
Time Frame: as for outcome 4
Population: Treatment-Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Extension Period: Ruxolitinib Cream 1.5% BID | Treatment-Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 37 | 14
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 52 + 30 days)
Description: Treatment-emergent adverse events (TEAEs): AEs reported for the first time or the worsening of a pre-existing event after the first application of study drug. For the Double-Blind Period, TEAEs are reported for members of the Safety Population: all participants who applied ruxolitinib cream or vehicle cream at least once. For the Treatment-Extension (TE) Period, TEAEs are reported for the TE Evaluable Population: all participants who applied ruxolitinib cream at least once in the TE Period.
Groups:
- Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib cream during the Double-Blind Treatment Period and the Treatment-Extension Period. Participants applied ruxolitinib 1.5% cream BID for 24 weeks. Participants who completed the Week 24 assessments with no safety concerns could continue into the 28-week Treatment-Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-Blind Period continued to apply ruxolitinib cream 1.5% BID for an additional 28 weeks in the Treatment-Extension Period. Participants who applied vehicle cream BID during the Double-Blind Period applied ruxolitinib cream 1.5% BID for 28 weeks in the Treatment-Extension Period.
- Vehicle Cream BID: Participants applied matching vehicle cream twice a day (BID) for 24 weeks in the Double-Blind Period.
Arm/Group | Ruxolitinib Cream 1.5% BID | Vehicle Cream BID
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/19
Other Adverse Events (participants affected / at risk) | 10/55 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Cream 1.5% BID (N=55) | Vehicle Cream BID (N=19)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Cream 1.5% BID (N=55) | Vehicle Cream BID (N=19)
Application site exfoliation (General disorders) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 9 (9) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT04896385/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04896385/SAP_001.pdf